CLINICAL TRIAL: NCT06631989
Title: A Phase I/II Multicenter, Open Label, Single-arm Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of WSD0922-FU in the Treatment of Advanced Non-small Cell Lung Cancer
Brief Title: A Study to Assess the Efficacy and Safety of WSD0922-FU in Patients With EGFRm+ Advanced Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wayshine Biopharm, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WSD0922-102
Record Dates: First submitted 2024-08-25; First posted 2024-10-08 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: EGFR Mutation Positive Advanced Non-Small Cell Lung Cancer
Keywords: NSCLC; EGFR; C797S; BM

STUDY DESIGN:
Intervention Model Description: Part A (Dose escalation and expansion study) ; Part B (single-arm extension study).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose escalation (WSD0922-FU) (Experimental): Patients receive WSD0922-FU PO QD on C0D1 to C0D3, then BID on C1D1 to C1D21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, MRI, and blood sample collection on study.
  Interventions: Drug: WSD0922-FU
- Dose expansion (WSD0922-FU) (Experimental): Patients receive WSD0922-FU PO BID on C1D1 to C1D21 using dosage selected from Dose escalation. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, MRI, and blood sample collection on study.
  Interventions: Drug: WSD0922-FU
- Dose extension (WSD0922-FU) (Experimental): Patients receive WSD0922-FU PO BID on C1D1 to C1D21 using RP2D. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, MRI, and blood sample collection on study.
  Interventions: Drug: WSD0922-FU

INTERVENTIONS:
Drug: WSD0922-FU — Procedure: Biospecimen Collection - blood samples Undergo collection of blood samples
  Procedure: Computed Tomography and/or Magnetic Resonance Imaging Undergo CT and/or MRI
  Drug: WSD0922-FU Given PO
  Other Names: WSD0922

SUMMARY:
This study is a multicenter, open label, single-arm phase I/II clinical trial of WSD0922-FU for patients with locally advanced or metastatic non-small cell lung cancer whose disease has progressed with thrid-generation EGFR-TKI .

DETAILED DESCRIPTION:
WSD0922-FU is a potent reversible inhibitor of both the single EGFRm+ and dual EGFRm+/C797S+ receptor forms of EGFR with selectivity margin over wild-type EGFR. This study aims to explore the safety, tolerability, pharmacokinetic characteristics and efficacy of WSD0922-FU in patients with non-small cell lung cancer (NSCLC) with C797S mutation after first-line third-generation EGFR-TKI resistance.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old (including the threshold value), gender is not limited;
* Locally advanced or metastatic NSCLC confirmed by pathology;
* Patients who have been genetically tested to carry EGFR sensitive mutations;
* Blood samples must be provided for testing and must be taken during or after disease progression following the last EGFR TKI inhibitor treatment;
* Must have a minimum life expectancy of >= 3 months;
* At least one measurable tumor lesion according to RECIST version 1.1; Previous radiotherapy-treated lesions cannot be used as target lesions unless imaging studies show clear progression of the lesions.
* Physical Status (ECOG PS) score was 0-1;
* Have full organ function;
* Eligible patients (male and female) who are fertile must agree to use a reliable contraceptive method ;
* Subjects are required to give informed consent to this study before the experiment and sign a written informed consent voluntarily.

Exclusion Criteria:

* Received chemotherapy, radiotherapy, biological therapy, targeted therapy, endocrine therapy, immunotherapy, or other anti-tumor drug treatments within 4 weeks before the first administration of the study drug.
* Have previously received more than one EGFR-TKI inhibitor;
* Received other unlisted clinical study drugs or treatments within 4 weeks before the first administration.
* Received major organ surgery (excluding puncture biopsy) or significant trauma within 4 weeks before the first administration, or require elective surgery during the trial period.
* Used strong CYP3A4 inhibitors or strong CYP3A4 inducers within 7 days before the first use of the study drug.
* Known active brain metastasis or progression evidence.
* Other primary malignant tumors within 2 years before the first administration of the study drug.
* Adverse reactions from previous anti-tumor treatments have not recovered to NCI-CTCAE v5.0 grade ≤1 (except for toxicities judged by the researcher to have no safety risks, such as hair loss, grade 2 peripheral neurotoxicity, and stable thyroid function after hormone replacement therapy).
* Skin/pressure ulcers, chronic leg ulcers, known active gastric ulcers, or non-healing wounds.
* History of severe allergies, or allergies to any active or inactive ingredients of the study drug;
* Severe infections requiring intravenous antibiotic infusion or hospitalization at the time of screening; or uncontrollable active infections within 4 weeks before administration;
* Known active or suspected autoimmune diseases; or known active ocular diseases (such as active wet age-related macular degeneration, diabetic retinopathy with macular edema);
* Human immunodeficiency virus (HIV) (HIV1/2 antibody) positive, syphilis spirochete antibody positive .
* Patients with interstitial lung disease.
* History of severe cardiovascular diseases.
* Unable to orally swallow medication, or there is a condition that significantly affects gastrointestinal absorption as judged by the researcher;
* Clinical intervention is required for pleural effusion, ascites (excluding subjects who do not need drainage and have been stable for more than 2 weeks after drainage).
* Known alcohol or drug dependence.
* Mental disorders or poor compliance;
* Pregnant or lactating women;
* The investigator believes that the subject has other reasons that make them unsuitable for participating in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR by IRC | every 6 weeks, up to 1 year
  proportion of patients with a best overall response of complete response or partial response
PartA: To evaluate the safety of WSD0922-FU in patients with NSCLC | 8 months
  Safety (incidence and severity of adverse events [AE])
PartA: To evaluate the tolerability of WSD0922-FU in patients with NSCLC | 8 months
  Incidence and quantity of dose-limiting toxicity (DLT)
PartA: To evaluate the Maximum Tolerated Dose (MTD) of WSD0922-FU in patients with NSCLC | 8 months
  Incidence of Dose-Limiting Toxicities (DLTs)
PartA: Recommended Phase II Dose (RP2D) of WSD0922-FU in patients with NSCLC | 8 months
  Recommended Phase II Dose (RP2D)

SECONDARY OUTCOMES:
PK exposure parameter: Maximum Plasma Concentration (Cmax) | 12 months
  Maximum Plasma Concentration (Cmax)
PK exposure parameter: Time To Maximum Plasma Concentration (Tmax) | 12 months
  Time To Maximum Plasma Concentration (Tmax)
PK exposure parameter: Area Under The Plasma Concentration-Time Curve From Time Zero To Time With Last Measurable Concentration (AUC0-t) | 12 months
  Area Under The Plasma Concentration-Time Curve From Time Zero To Time With Last Measurable Concentration (AUC0-t)
PK exposure parameter: Area Under The Plasma Concentration-Time Curve From Time Zero To Infinity (AUC0-∞) | 12 months
  Area Under The Plasma Concentration-Time Curve From Time Zero To Infinity (AUC0-∞)
PK exposure parameter: Terminal Elimination Half-Life (t½) | 12 months
  Terminal Elimination Half-Life (t½)
PK exposure parameter: Apparent Terminal Elimination Rate Constant (λz) | 12 months
  Apparent Terminal Elimination Rate Constant (λz)
PK exposure parameter: Apparent Clearance (CL) | 12 months
  Apparent Clearance (CL)
PK exposure parameter: Apparent volume of distribution (Vd) | 12 months
  Apparent volume of distribution (Vd)
PK exposure parameter: Mean Residence Time (MRT) | 12 months
  Mean Residence Time (MRT)
Steady state pharmacokinetic parameter: Area Under the Steady-State Concentration-Time Curve（AUCss） | 12 months
  Area Under the Steady-State Concentration-Time Curve（AUCss）
Steady state pharmacokinetic parameter: Area Under the Steady-State Concentration-Time Curve from 0 to Infinity（AUC0-∞,ss） | 12 months
  Area Under the Steady-State Concentration-Time Curve from 0 to Infinity（AUC0-∞,ss）
Steady state pharmacokinetic parameter: Area Under the Steady-State Concentration-Time Curve from 0 to Time t （AUC0-t,ss） | 12 months
  Area Under the Steady-State Concentration-Time Curve from 0 to Time t （AUC0-t,ss）
Steady state pharmacokinetic parameter: Average Steady-State Concentration（Cav） | 12 months
  Average Steady-State Concentration（Cav）
Steady state pharmacokinetic parameter: Steady-State Clearance（CLss） | 12 months
  Steady-State Clearance（CLss）
PK exposure parameter :Maximum Steady-State Concentration（Cmax,ss） | 12 months
  Maximum Steady-State Concentration（Cmax,ss）
PK exposure parameter : Minimum Steady-State Concentration（Cmin,ss） | 12 months
  Minimum Steady-State Concentration（Cmin,ss）
PK exposure parameter : Trough Concentration（Ctrough） | 12 months
  Trough Concentration（Ctrough）
PK exposure parameter : Fluctuation Degree（DF） | 12 months
  Fluctuation Degree（DF）
PK exposure parameter : Accumulation Ratio（Ra） | 12 months
  Accumulation Ratio（Ra）
PK exposure parameter : Time to Maximum Concentration at Steady State（Tmax,ss） | 12 months
  Time to Maximum Concentration at Steady State（Tmax,ss）
PK exposure parameter : Volume of Distribution Calculated from the Terminal Elimination Phase（Vz） | 12 months
  Volume of Distribution Calculated from the Terminal Elimination Phase（Vz）
To evaluate the safety of WSD0922-FU in patients with advanced non-small cell lung cancer | 12 months
  Treatment-Emergent Adverse Events (TEAEs), Treatment-Related Adverse Events (TRAEs)
ORR by investigators | every 6 week, up to 12 months
  proportion of patients with a best overall response of complete response or partial response
Disease Control Rate (DCR) | every 6 weeks, up to12 months
  the percentage of patients who have a best overall response of CR or PR or SD
Duration of Response (DoR) | every 6 weeks, up to 12 months
  proportion of patients with the time from the date of first documented response until the date of documented progression or death in the absence of disease progression
PFS | every 6 weeks, up to 12 months
  proportion of patients with the time from randomization until the date of objective disease progression or death
OS | 24 months
  proportion of patients with the time from randomization until the date of objective disease progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, MD, Principal Investigator — Shanghai East Hospital
Locations (12):
- China (12):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - He'nan Cancer Hospital, Zhengzhou, Henan
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Sichuan Provincial Cancer Hospital, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No